CLINICAL TRIAL: NCT05563038
Title: Scrambler Therapy for Post-Stroke Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00323440
Record Dates: First submitted 2022-09-28; First posted 2022-10-03 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Post Stroke Pain

STUDY DESIGN:
Intervention Model Description: Scrambler Group and Non-scrambler group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Scrambler Therapy (Active Comparator): Using Scrambler Therapy for Post Stroke Pain all participants will either undergo either 5 or 10 treatments using Scrambler Therapy. The number of treatments will be decided by a randomization process.
  Interventions: Device: Scrambler Therapy for Post Stroke Pain

INTERVENTIONS:
Device: Scrambler Therapy for Post Stroke Pain — All participants will either undergo either 5 or 10 treatments using Scrambler Therapy. The number of treatments will be decided by a randomization process.

SUMMARY:
The Investigators will enroll patients who have had a stroke and are experiencing post-stroke pain secondary to their infarct and disruption of the sensory system in a research study to compare the effectiveness of Scrambler Therapy to traditional pharmacologic therapies.

DETAILED DESCRIPTION:
Participants will work with the provider to decide which method of treatment they prefer and will then be followed regularly using standardized pain scores over the next year.

Those undergoing ST will undergo 5-10 sessions while those treated with medical therapy will undergo titration of medication as per typical standard of care. The investigators will compare both maximal pain relief achieved and duration achieved between groups.

prospectively enroll a consecutive series of patients presenting to clinic with post-stroke pain syndromes following either an ischemic infarct or intracranial hemorrhage. Patients will be included in the study if they are at least one month post-stroke (but can be chronic) and have pain in an area attributable to the location of their lesion (ie contralateral to a lesion involving the thalamus or sensory cortex). At their clinic visit, potential treatments: Scrambler Therapy or pharmacological treatment, will be discussed with each patient. Patients will not be excluded if they are currently taking or have taken pain medications in the past, though these variables will be factored into the analysis. Through shared decision making, the investigator along with the patients input will decide on ST versus medical management. Participants will consent to being followed for pain control over the following year of therapy to enable comparison of ST to standard medical therapy.

All patients will begin by rating their current pain on the Numerical Rating Scale (NRS) from 0-10.

Patients undergoing treatment by Scrambler Therapy will begin by describing the areas and levels of pain along the Numerical Rating Scale (NRS) from 0-10. The dermatomes of the areas of pain will be examined by going up and down the dermatome as shown on a dermatome map, and the electrode of the Scrambler machine will be placed at the site where pain is initiated and approximately 10 centimeters above it. The Scrambler machine will then be started and turned on until patients feel a "tingling" sensation that is not painful. For approximately 45 minutes, the Scrambler machine will run while a team member watches over the patient, adjusting the levels only if the patient no longer feels the tingling sensation.

After the Scrambler treatment, patients will again be asked to describe the areas and levels of pain using the NRS. Each patient undergoing Scrambler Therapy will undergo this process for 5 consecutive days, following the same procedure every day of treatment. After completion of treatment, participants will be asked to complete monthly ratings of their pain for three months, and to follow-up in clinic at 3-6 month intervals (standard of care).

While the mechanism of action of ST in treating CNS pain is unknown, thalamocortical dysrhythmia (TD) is one mechanism hypothesized to underlie post-stroke pain that may be affected by the neuromodulation. The thalamus serves as a connection hub between cortical sensory regions and areas of pain perception. Prior work suggests that with TD there is increased low frequency (beta and theta) bursting within dorsal anterior cingulate cortex (dACC) and abnormalities within the default mode, central executive, and salience networks. These abnormalities are observed in patients with chronic pain. We hypothesize the same is true for post-stroke pain and that ST modulates the aberrant thalamocortical signaling, reducing maladaptive beta-band activity within the dACC for patients with significant reductions in pain after treatment. In this proposal, we will build upon our established infrastructure to collect neuroimaging data from 100 patients who experience post-stroke pain, each undergoing 5 sessions of ST. Pain scores will be recorded at baseline and before and after each session. Magnetoencephalography (MEG) will be performed at baseline, and post- treatments #1 and #5 to investigate for signs of thalamocortical dysrhythmia by comparing neural responses from this cohort to those of a similar, previously-collected cohort with no post-stroke pain. We will then determine the changes in neural activity associated with favorable treatment response (>50% reduction in pain score at visit #5) among treated individuals, and evaluate whether neural changes following visit #1 combined with baseline variables are sufficient to predict overall treatment response. The proposal is built around the following specific aims:

Aim 1: Investigate the role of TD in post-stroke pain by evaluating neuroimaging features present in symptomatic patients compared to controls. Spectral and functional connectivity analyses will be performed to evaluate whole brain differences at baseline between groups with specific focus on 1) low frequency activity within the dACC and 2) differences within the default mode, central executive, and salience networks.

Hypothesis 1: Affected patients will show high levels of beta activity within the dACC compared to controls without pain supporting thalamocortical dysrhythmia as an underlying mechanism.

Aim 2: Determine the neuroimaging patterns associated with favorable treatment response in patients treated with ST. Similar analyses will also be performed at each time point (baseline, post-#1, -#5) to evaluate differences between patients treated with ST who show significant response to treatment versus non-responders.

Hypothesis 2: 1) High levels of beta activity will be present within the dACC at baseline for all patients, but resolve in patients with >50% reduction in pain scores post-visit #5, and 2) patients with the highest baseline levels of beta activity within the dACC will see the greatest absolute decrease in pain scores over time.

Aim 3: Create a multivariable predictive model to guide future treatment. Differences in neural activity observed post-visit #1 for responders versus non-responders, along with demographic information, stroke characteristics, and additional treatment variables will be used in regression analyses to create a multivariable model of factors associated with favorable treatment response in a training cohort. ROC analysis will be used to determine the sensitivity and specificity of the model, which will be internally validated for in a smaller test cohort.

Hypothesis 3: 1) Patients with the greatest decrease in beta activity as a result of treatment #1 will see the greatest absolute reduction in pain post-visit #5. 2) Strokes involving either of the bilateral thalami will be less likely to result in >50% reduction in pain independent of treatment duration, and concurrent use of medications (SNRIs, TCAs, or antiepileptics) will improve the efficacy of ST.

Using MEG to better understand the underlying neural mechanisms responsible for post-stroke pain and treatment response will allow us to better predict response to therapy and individualize treatment paradigms in future clinical trials based on biomarkers to maximize response, leading to decreased post-stroke morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over the age of 18 with ischemic or hemorrhagic stroke seen on imaging and a positive finding for pain in the area(s) affected by their stroke location will be included.
* The patients must be at least one month post-stroke but can otherwise enroll at any point.

Exclusion Criteria:

* Patients with TIA
* Patients with no evidence of stroke on MRI
* Patients with implantable devices such as pacemakers, defibrillators, spinal cord stimulators
* Patients with history of myocardial infarction in the past 6 months
* Patients with uncontrolled epilepsy
* Patients with symptomatic brain metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Reduction in post stroke pain | 6 months
  At least a 50% reduction in post stroke pain

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Merbach, MNP, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No